CLINICAL TRIAL: NCT02056132
Title: Exhaled Breath Condensate for Evaluation of Lung Infections and Exacerbations in Patient With Cystic Fibrosis.
Brief Title: Breath Condensate Study in Patients With Cystic Fibrosis.
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201200137
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Exhaled breath condensate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis patients.: Patients with Cystic Fibrosis. Results of Exhaled Breath Condensate lab.
  Interventions: Other: Exhaled Breath Condensate
- Control Subjects: Individuals without Cystic Fibrosis or signs of current respiratory infection. Results of Exhaled Breath Condensate lab.
  Interventions: Other: Exhaled Breath Condensate

INTERVENTIONS:
Other: Exhaled Breath Condensate — Lab results of Exhaled Breath Condensate

SUMMARY:
There is an urgent need for a noninvasive method to diagnose bronchial infections and exacerbations in patients with Cystic Fibrosis (CF). The current method to diagnosed infections involves either collecting a sputum sample or obtaining a bronchoalveolar lavage (BAL). However, some patients cannot produce sputum. At the same time the decision of when a patient has an exacerbation continues to be very subjective. In this exploratory study, we propose a new, noninvasive method to diagnose bronchial infections and to evaluate possible markers of inflammation that can assist in a noninvasive way in the determination of exacerbations.

DETAILED DESCRIPTION:
We hypothesize that it is possible to recover microbial products causing infections in Exhaled Breath Condensate (EBC) samples as well as to measure markers of inflammation like Interleukin (IL)-8, Leukotriene B4 (LTB4), Interleukin IL-6, Interleukin IL-1B, Tumor Necrosis Factor alpha, as well as proteases like neutrophil elastase, matrix metalloproteinase 2 and 9 and antiproteases like secretory leukoprotease inhibitor (SLPI), alpha one antitrypsin and tissue inhibitor of metalloproteinase-1 (TIMP-1). As a way to compare our findings to systemic inflammation we will also measure C-reactive protein in serum.

20 patients with cystic fibrosis who have chronic bronchial infection and 20 controls will be recruited. Their exhaled breath condensate and sputum samples will be collected and analyzed for the presence of bacteria through traditional, molecular and nuclear acid amplification methods as well as Pyrosequencing analysis. We will also measure the above markers of inflammation and follow the CF patients for the following year so we can continue to collect exhaled breath condensate when they have an exacerbation and are admitted to the hospital as well as after treatment for the exacerbation. We will correlate these markers with patient's clinical features including pulmonary function test, Body max index, CF pathogens, and CF genotype. If our hypothesis turns out to be true it will open up a possibility for a new noninvasive diagnostic and follow up method that will benefit cystic fibrosis patients.

2. Hypothesis & Specific Aims:

A. Microbial products can be recovered from exhaled breath condensate. B. That these microbial products recovered from exhaled breath correlate with that recovered from sputum C. Markers of inflammation can be recovered from exhale breath condensate.

ELIGIBILITY:
Inclusion Criteria:

Any patient with Cystic Fibrosis (CF) in the age range 18-65 years who is known to be chronically infected in their respiratory tract will be eligible as cases. Any other patient or healthy subject in the age range 18-65 years who is not infected with Pseudomonas in their respiratory tract will be eligible as controls.

Exclusion Criteria:

Any study subject, who cannot co-operate with the study, cannot co-ordinate breathing or cannot breathe through a mouthpiece.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with Cystic Fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
correlation of EBC finding with exacerbations. | 1 year

SECONDARY OUTCOMES:
ability to identify common airway pathogens on EBC. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Lascano, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States